CLINICAL TRIAL: NCT07002164
Title: Trial of IMmediate Invasive Versus Delayed Coronary ANGiography in Non-ST-Segment Elevation Myocardial Infarction Complicated by Acute Decompensated Heart Failure: The TIMING-AHF Trial
Brief Title: Timing of Coronary Angiography in NSTEMI Complicated by Acute HF
Acronym: TIMING-AHF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Min Chul Kim, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2025-100
Record Dates: First submitted 2025-05-17; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction (MI); Heart Failure
Keywords: Non-ST-segment elevation myocardial infarction; Acute decompensated heart failure; Coronary angiography; Timing
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate coronary angiography within 2 hours after diagnosis of non-ST-segment elevation myocardial (Experimental): Coronary angiography will be performed within 2 hours after diagnosis of non-ST-segment elevation myocardial infarction.
  Interventions: Procedure: Immediate coronary angiography
- Delayed coronary angiography after stabilization of acute decompensated heart failure (Active Comparator): Coronary angiography will be performed after disappearance of symptoms and signs of acute decompensated heart failure.
  Interventions: Procedure: Delayed coronary angiography

INTERVENTIONS:
Procedure: Immediate coronary angiography — Immediate coronary angiography ≤2 hours after randomization
  Arms: Immediate coronary angiography within 2 hours after diagnosis of non-ST-segment elevation myocardial
Procedure: Delayed coronary angiography — Delayed coronary angiography after stabilization
  Arms: Delayed coronary angiography after stabilization of acute decompensated heart failure

SUMMARY:
Study objectives:

To determine the optimal timing of coronary angiography (CAG) in patients with non-ST-segment elevation myocardial infarction (NSTEMI) complicated by acute decompensated heart failure (AHF). The primary objective of this trial is to test the hypothesis that immediate CAG ≤2 hours after establishment of NSTEMI diagnosis would result in a significant reduction in primary composite outcome of death from any cause, non-fatal myocardial infarction (MI), or hospitalization for heart failure (HF) at 12 months after randomization as compared with delayed CAG after stabilization.

Study hypothesis:

Immediate CAG ≤2 hours after establishment of NSTEMI diagnosis would result in a significant reduction in primary composite outcome of death from any cause, non-fatal myocardial infarction (MI), or hospitalization for heart failure (HF) at 12 months after randomization as compared with delayed CAG after stabilization.

Background:

Although current guidelines recommend early CAG within 2 hours for patients with NSTEMI complicated by AHF, many patients with NSTEMI complicated by AHF did not receive early CAG. However, no randomized clinical trials have evaluated the optimal timing of CAG in patients with NSTEMI complicated by AHF. Therefore, the investigators aimed to perform a prospective, investigator-initiated, open-label, muilticenter trial to compare the efficacy and safety between immediate CAG (CAG <2 hours after establishment of NSTEMI diagnosis) and delayed CAG after stabilization (i.e. improved dyspnea and disappearance of pulmonary congestion) in participants with NSTEMI complicated by AHF.

Study procedure:

Following the establishment of NSTEMI diagnosis, participants fulfilling the eligibility criteria will be randomized at a ratio of 1:1 to immediate CAG ≤2 hours after randomization or delayed CAG after stabilization on another day during hospitalization.

DETAILED DESCRIPTION:
Acute decompensated heart failure (AHF) is frequently encountered in patients with non-ST-segment elevation myocardial infarction (NSTEMI), and it is known to be associated with worse clinical outcomes that those without heart failure (HF). Although current guidelines recommend immediate invasive strategy for patients with NSTEMI complicated by AHF, its evidence is lack. It is difficult to decide whether to perform early coronary angiography (CAG) according to the guidelines in these high-risk patients due to the risk of procedural complications. Furthermore, the most of randomized trials regarding the timing of CAG in non-ST-segment elevation acute coronary syndrome (NSTE-ACS) have excluded these patients, therefore, there is lack of evidence for performing immediate CAG in such cases. In clinical practice, many patients with NSTEMI complicated by AHF did not receive early CAG. There are only two observational studies which investigated this issue. In the Korean nationwide registry data, a total of 1,027 patients with NSTEMI complicated by AHF were analyzed, and 14.5% among study population underwent early CAG within 2 hours according to the guidelines. All-cause mortality at 12 months was not significantly different irrespective of CAG timing. In other single-center study, early CAG <24 hours was associated with a lower risk of adverse cardiac outcomes compared with delayed CAG ≥24 hours after admission.

Several studies have demonstrated improved clinical outcomes in high-risk patients with NSTE-ACS undergoing early CAG, whereas others have found no significant differences in clinical outcomes. Randomized clinical trials, such as SISCA, ISAR-COOL, RIDDLE-NSTEMI and EARLY, have demonstrated the advantages of early CAG compared to delayed invasive approach (i.e. CAG after stabilization) in high-risk patients with NSTE-ACS. The other trials regarding this issue have failed to show the superiority of early CAG over delayed invasive approach. However, no randomized clinical trials have evaluated the optimal timing of CAG in patients with NSTEMI complicated by AHF.

Therefore, the investigators aimed to perform a prospective, investigator-initiated, open-label, muilticenter trial to compare the efficacy and safety between immediate CAG (CAG <2 hours after establishment of NSTEMI diagnosis) and delayed CAG after stabilization (i.e. improved dyspnea and disappearance of pulmonary congestion) in participants with NSTEMI complicated by AHF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* Non-ST-segment elevation myocardial infarction
* New-onset or worsening of dyspnea (New York Heart Association class ≥2)
* Pulmonary congestion
* Patient's or guardian's consent after understanding the study

Exclusion Criteria:

* Cardiogenic shock at initial presentation
* ST-segment elevation myocardial infarction

  * ST-segment elevation ≥0.1 mV in at least 2 contiguous leads, or
  * New onset left bundle branch block
  * Posterior wall myocardial infarction
* Refractory angina
* Life threatening ventricular arrhythmias
* Life expectancy <1 year
* Apparently non-ischemic cause of HF
* Pregnancy and lactation
* History of coronary artery bypass grafting (CABG), or planned CABG
* Patient's refusal to participate in study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
A cumulative incidence rate of all-cause death, non-fatal myocardial infarction (MI), or hospitalization for heart failure (HF) | 1 year

SECONDARY OUTCOMES:
A cumulative incidence rate of all-cause death, non-fatal MI, or hospitalization for HF | 1, 6, 24, 36 months
All-cause death | 1, 6, 12, 24, 36 months
Non-fatal MI | 1, 6, 12, 24, 36 months
Hospitalization for HF | 1, 6, 12, 24, 36 months
Cardiovascular death | 1, 6, 12, 24, 36 months
Recurrent ischemia | 1, 6, 12, 24, 36 months
  Recurrent ischemia is defined as repeated episodes of ischemic symptoms needing emergent coronary angiography with any of the following signs:
  * Electrocardiographic changes indicating myocardial ischemia
  * Ventricular arrhythmias
  * New-onset pulmonary edema
  * Cardiogenic shock
All unplanned revascularization | 1, 6, 12, 24, 36 months
Definite or probable stent thrombosis | 1, 6, 12, 24, 36 months
Stroke | 1, 6, 12, 24, 36 months
Major bleeding by Bleeding Academic Research Consortium | 1, 6, 12, 24, 36 months
Acute kidney injury (AKI) and AKI requiring renal replacement therapy | Up to 7 days
In-hospital death rate from any cause | Up to 30 days
In-hospital death rate from cardiovascular cause | Up to 30 days

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Gyeongsang National University Changwon Hospital, Changwon
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeongnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gwangju Veterans Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Dong-A University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Koera University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - St. Carollo General Hospital, Suncheon
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No